CLINICAL TRIAL: NCT06755359
Title: A Safety Study of Intratumoral Diffusing Alpha Radiation Emitters With Chemotherapy for the Treatment of Locally Advanced Pancreatic Cancer
Brief Title: Alpha Radiation Emitters Device (DaRT) for the Treatment of Locally Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-PANC-04
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; Locally Advanced Pancreatic Cancer
Keywords: Alpha radiation; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — Radioactive sources named Alpha DaRT sources: Ra - 224 coated onto titanium tubes inserted into the tumor.

SUMMARY:
A unique approach for cancer treatment including radioactive sources named Alpha DaRT sources: Ra - 224 coated onto stainless steel tubes inserted into the tumor for the treatment of Locally Advanced Pancreatic Cancer .

DETAILED DESCRIPTION:
This study will be a prospective, interventional, open label, single arm, multiple center study.

Patients who have been previously treated with 8 - 12 cycles of mFOLFIRINOX will undergo DaRT insertion, with the goal of making their tumor resectable. Three (3) days after DaRT insertion, patients will begin taking Capecitabine for 2 months. Every 2 months after DaRT insertion, the patient will be assessed to determine if their tumor is surgically resectable, if they should continue with therapy, or if they should pause therapy. The trial will end 12 months after DaRT insertion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven locally advanced pancreatic adenocarcinoma
* Target lesion is technically amenable for Alpha DaRT sources implantation.
* Measurable lesion per RECIST (version 1.1) criteria
* Stable disease or tumor response per RECIST (version 1.1) criteria compared to before initiation of mFOLFIRINOX
* Lesion size ≤ 5 cm in the longest diameter
* Interstitial radiation indication validated by a multidisciplinary team which includes an oncologist, a radiation oncologist, radiologist, gastroenterologist and a surgeon specialized in pancreatic oncology in the case that a surgical emergency occurs during the procedure
* Patients have received 8 - 12 cycles of mFOLFIRINOX
* ECOG Performance Status Scale 0 - 1
* Life expectancy is more than 6 months
* WBC ≥ 3500/µl, granulocyte ≥ 1500/µl
* Platelet count ≥60,000/µl
* Creatinine ≤1.9 mg/dL
* AST and ALT ≤ 2.5 X upper limit of normal (ULN)
* INR < 1.4 for patients not on Warfarin
* Age ≥18 years old
* Subjects are willing and able to sign an informed consent form
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test before the Ra-224 implantation and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after initiation of Alpha DaRT therapy
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after DaRT insertion.

Exclusion Criteria:

* Concomitant immunotherapy within the past 4 weeks.
* Patients with metastatic disease
* Borderline unresectable pancreatic cancer, and/or cases fit for surgical exploration unless patient refuses surgery.
* Known hypersensitivity to any of the components of the treatment.
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, low risk prostate cancer, or in situ cervical cancer.
* Patient requires treatment not specified in this protocol which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT.
* Patients do not agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Breastfeeding women or women of childbearing potential unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 3 months after RT.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety - Serious adverse events | from Day 0 , up to 12 months
  Safety will be determined according to the overall incidence of device related SAEs with severity graded according to CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Efficacy - tumor response | Day 0 , up to 12 months
  to evaluate the efficacy of the Alpha DaRT sources in advanced pancreatic cancer patients with respect according to Objective tumor response rate according to RECIST 1.1
Efficacy - overall survival | Day 0 , up to 12 months
  to evaluate the efficacy of the Alpha DaRT sources in advanced pancreatic cancer patients with respect according to Overall survival
Efficacy - Progression-free survival | Day 0 , up to 12 months
  to evaluate the efficacy of the Alpha DaRT sources in advanced pancreatic cancer patients with respect according to - Progression-free survival
Efficacy - Percentage of R0/R1 resected patients | Day 0 , up to 12 months
  to evaluate the efficacy of the Alpha DaRT sources in advanced pancreatic cancer patients with respect according to Percentage of R0/R1 resected patients
Efficacy - percentage of patients with tumors that became surgically respectable after DaRT treatment | Day 0 , up to 12 months
  to evaluate the efficacy of the Alpha DaRT sources in advanced pancreatic cancer patients with respect according to percentage of patients with tumors that became surgically respectable after DaRT treatment

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU de Bordeaux, Bordeaux
  - Centre Jean PERRIN - Clermont-Ferrand, Clermont-Ferrand
  - Centre Georges François Leclerc Dijon, Dijon
  - CHU Grenoble Alpes, Grenoble
  - Hôpital Privé Mermoz - Lyon, Lyon
  - Marseille, Marseille
  - CHU Poitiers, Poitiers
  - Gustave Roussy Institute, Villejuif